CLINICAL TRIAL: NCT01296113
Title: Phase II Trial Evaluating the Efficacy and Safety of Carboplatin Plus Pemetrexed in Human Immunodeficiency Virus Positive (HIV+) Patients With Stage III (Not Amenable to Radiation or Inoperable) or Stage IV Nonsquamous Non Small Cell Lung Cancer
Brief Title: Chemotherapy for Lung Cancer in HIV-positive Patients
Acronym: CHIVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-1001
Record Dates: First submitted 2011-02-11; First posted 2011-02-15 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Non-small Cell Lung Cancer; Hiv-positive
Keywords: IFCT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; HIV Seropositivity | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Pemetrexed + Carboplatin
  On D1 of a 21-day cycle:
  * Pemetrexed 500 mg/m² IV in 10 minutes followed 30 minutes later by:
  * Carboplatin AUC 5 in 30 minutes in 100 ml sterile water or 5% glucose or physiological serum. The carboplatin dose will be calculated by the Calvert formula with a target AUC of 5 mg/mL.min as follows:
  Carboplatin dose in mg = 5 x (GFR + 25) GFR is estimated according to the MDRD equation for creatinine clearance
  • 4 cycles total

SUMMARY:
This is a phase II, multicenter, non-randomized, open-label study evaluating the combination of pemetrexed plus carboplatin in HIV-positive patients with lung cancer.

DETAILED DESCRIPTION:
The use of tritherapy in developed countries starting in 1996 led to a considerable reduction in AIDS mortality due to opportunistic infections and AIDS-defining cancers. However, increased life expectancies were accompanied by a diversification of the causes of death in HIV-infected individuals. In France between 2000 and 2005, non-AIDS-defining mortality rose from 53% to 64%: non-AIDS-defining cancers (apart from hepatocellular carcinoma) had the highest mortality rates, increasing from 11% to 17% in 2005, followed by liver disease (15% in 2005), cardiovascular disease (8% in 2005) and suicide (5%). Among all cancer-related deaths (AIDS- and non-AIDS-defining), the proportion due to non-AIDS-defining cancers (apart from hepatocellular carcinoma) increased from 38% to 50% and lung cancer (LC) accounted for 65% of deaths. Many epidemiological studies have demonstrated an elevated risk of LC in HIV-infected individuals HIV-positive subjects are younger at diagnosis of LC than the general population (45 versus 62 years). In the most recent studies, adenocarcinoma comprised 70% of cases. The prognosis of LC is worse in HIV-positive individuals. Some authors suggest that these poor outcomes may be related to interactions and additive toxicities of the cytotoxic and antiretroviral drugs. It is also likely that the disease is particularly aggressive. In the general population with a PS of 0 or 1 and under 70 years of age, bitherapy improves survival as compared to monotherapy. Survival is higher when the doublet comprises a platin. Since HIV-positive subjects with LC tend to be young, it is logical to offer them the best treatment which has demonstrated efficacy in the general population. In comparison to cisplatin, carboplatin causes less vomiting, nephrotoxicity and neurotoxicity. Survival is very slightly higher with cisplatin, but this comes at the cost of greater toxicity. Carboplatin is better tolerated in subjects with PS=2 or who are over 70 years of age

The HIV-positive population is specific in that:

* PS is more often altered but the subjects are young, which calls for a platin-based doublet.
* HAART is essential and its absorption should not be compromised by repeated vomiting which is more severe with cisplatin.
* Nephropathy occurs in 15-38% of cases; the causes are multifactorial and include the HIV virus itself and the antiretroviral drugs (Tenofovir®).
* Peripheral neuropathy is frequently related to HIV or to the antiretroviral treatments (especially didanosine or stavudine (2010 YENI report)).
* Premature ageing is seen in HIV-positive subjects; this exposes them to increased cardiovascular risk and a higher frequency of heart disease which can restrict the hyper-hydration required when using cisplatin.
* In 2010, virtually all patients are treated on an ambulatory basis whereas in the past they would have been hospitalized. Carboplatin is administered in the day hospital of all the centers, but not cisplatin.
* It is important to preserve an optimal quality of life during the first line of therapy in these patients whose life expectancy is such that very few will be eligible for a second round of therapy.

Scagliotti published a phase III trial comparing cisplatin plus pemetrexed with cisplatin plus gemcitabine in subjects < 70 years old with advanced-stage NSCLC. Overall survival was identical in both arms but the toxicity profile was in favor of the pemetrexed arm. The combination of first-line carboplatin plus pemetrexed has been evaluated in several phase II trials, particularly in subjects with a poor PS. In contrast to the taxanes or vinorelbine, for example, pemetrexed is not metabolized by CYP450, which facilitates its use in combination with protease inhibitors and NNRTI, which respectively inhibit or induce the CYP450 system.

Ancillary study BIO-IFCT-1001 will be made. Since the samples will be small, focus will be on the biomarkers associated with multiple or specific resistance to platinum salts or to pemetrexed, particularly those more specifically found in NSCLC of nonsquamous histology. Similarly, biomarkers for which IFCT pathologists have acquired an expertise will also be favored. This expertise mainly involves, on the one hand, detecting K-Ras mutations (15-25% of ADC) and RasSF1 methylation as well as TubIII expression by immunohistochemistry (IHC) and testing for mucosecretion by PAS diastase-resistant staining, and on the other hand, evaluating ERCC1 and/or MSH2 expression and thymidylate synthase (TS) expression by IHC.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC histologically (highly recommended) and/or cytologically confirmed, stage III (non-irradiable or inoperable) or stage IV (according to 2009 TNM classification), with other than predominantly squamous histology
* HIV seropositivity (previous or inaugural), irrespective of CD4 count or viral load
* Presence of at least one measurable lesion (RECIST v1.1)
* Subject having signed the informed consent form,
* Subject who, in the investigator's opinion, will be able to comply with the requirements and constraints of the study
* Age ≥ 18 years ≤ 75 years,
* WHO performance status: 0, 1 or 2
* Weight loss ≤ 10% of total body weight in the month before inclusion
* Estimated life expectancy ≥ 1 month,
* Covered by health insurance

Exclusion Criteria:

* Bronchial cancer already treated (other than endoscopic deobstruction)
* Cancer which is amenable to surgery or radiation (curative),
* Squamous cell lung cancer or mixed small cell and non-small cell cancer, small cell lung cancer
* Creatinine clearance (MDRD) < 45 mL/min
* Severe hypersensitivity to any of the study products or excipients
* Severe disease or uncontrolled systemic disease (unstable or decompensated respiratory disease, cardiac, hepatic or renal disease, uncontrolled opportunistic infection)
* Significant abnormality in CBC-platelets (Hb <9 g/dL, PNN <1500 / mm3, platelets < 100,000 / mm3)
* Significant abnormality in liver tests (AST, ALT > 3x ULN, and <5 in case of liver metastases),
* Women of childbearing age without effective contraception; pregnant or breastfeeding women
* Subject who cannot take vitamin B12, folic acid or corticosteroids
* Diffuse interstitial pneumonia
* Any geographical situation or psychological condition that precludes full understanding and compliance with the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-05; Primary Completion 2016-01 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Disease-Control rate after 4 cycles | 3-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Armelle LAVOLE, MD, Principal Investigator — AP-HP, Hôpital Tenon
Locations (40):
- France (40):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Annemasse - CH, Ambilly
  - Annecy - CH, Annecy
  - Avignon - CH, Avignon
  - CH de la Côte Basque, Bayonne
  - CHU Besancon - Pneumologie, Besançon
  - Caen - CHU Côte de Nacre, Caen
  - CH Cahors, Cahors
  - CHU, Clermont-Ferrand
  - CH, Colmar
  - CH Compiègne - Pneumologie, Compiègne
  - Créteil - CHI, Créteil
  - CHU Grenoble - pneumologie, Grenoble
  - Le Mans - Centre Hospitalier, Le Mans
  - CH, Longjumeau
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Louis Pradel, Lyon
  - APHM - Hôpital Nord, Marseille
  - Montpellier - CHRU, Montpellier
  - Nevers - CH, Nevers
  - Centre Antoine Lacassagne, Nice
  - CHR d'Orléans La Source, Orléans
  - APHP - Hopital Tenon - Pneumologie, Paris
  - GH Paris Saint-Joseph, Paris
  - Hôpital Saint Antoine, Paris
  - Paris - Pitié-salpêtrière, Paris
  - Pau - CH, Pau
  - Centre François Magendie - hôpital du Haut-Lévèque, Pessac
  - HCL - Lyon Sud (Pneumologie), Pierre-Bénite
  - Reims - CHU, Reims
  - Rennes - CHU, Rennes
  - Saint Brieuc - CHG, Saint-Brieuc
  - NHC - Pneumologie, Strasbourg
  - Suresnes - Hopital Foch, Suresnes
  - Thonon les bains - CH, Thonon-les-Bains
  - Toulon - CHI, Toulon
  - CHU Toulouse - Pneumologie, Toulouse
  - Tourcoing - CH, Tourcoing
  - Tours - CHU, Tours
  - CH Valence, Valence

REFERENCES:
- [Background] Lavole A, Chouaid C, Baudrin L, Wislez M, Raguin G, Pialoux G, Girard PM, Milleron B, Cadranel J. Effect of highly active antiretroviral therapy on survival of HIV infected patients with non-small-cell lung cancer. Lung Cancer. 2009 Sep;65(3):345-50. doi: 10.1016/j.lungcan.2008.11.018. Epub 2009 Jan 9. PMID 19135758
- [Result] Lavole A, Greillier L, Mazieres J, Monnet I, Kiakouama-Maleka L, Quantin X, Spano JP, Lena H, Fraisse P, Janicot H, Audigier-Valette C, Langlais A, Morin F, Makinson A, Cadranel J; French Cooperative Thoracic Intergroup (IFCT). First-line carboplatin plus pemetrexed with pemetrexed maintenance in HIV-positive patients with advanced non-squamous non-small cell lung cancer: the phase II IFCT-1001 CHIVA trial. Eur Respir J. 2020 Aug 27;56(2):1902066. doi: 10.1183/13993003.02066-2019. Print 2020 Aug. PMID 32444410
- See also: IFCT official website — http://www.ifct.fr